CLINICAL TRIAL: NCT00847418
Title: Pharmacokinetics and Pharmacodynamics of Nasally Applied Esketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Qualified Person, Stefanie Deuster, PhD., Hospital Pharmacy, University Hospital Basel, Switzerland.
Other Study IDs: EKBB 351/08, 2009DR1015
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Pain
Keywords: pharmacokinetics; ketamine; Anesthetics, Dissociative
MeSH Terms: conditions — Pain

ARMS (1):
- Esketamine (Experimental)
  Interventions: Drug: esketamine hydrochloride

INTERVENTIONS:
Drug: esketamine hydrochloride

SUMMARY:
The purpose of this study is the determination of blood concentration and the effectiveness of esketamine after nasal application.

ELIGIBILITY:
Inclusion Criteria:

* male
* age ≥18 years ≤ 45 years
* healthy
* non-smoking
* BMI 18-27

Exclusion Criteria:

* abuse of drugs
* known or supposed hypersensitivity and/or contraindication against ketamine or additives
* participation of another clinical study within the last 30 days
* chronic obstructed nose breathing or nasal polyps
* dug allergy
* blood donation within the last two months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2009-02; Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, MD, Principal Investigator — Clinical Pharmacology and Toxicology, University Hospital Basel
Locations (1):
- Clinical Research Center, University Hospital Basel, Basel, Canton of Basel-City, Switzerland